CLINICAL TRIAL: NCT01218464
Title: Phase Ⅰ/Ⅱ Study of Human Umbilical Cord Derived Mesenchymal Stem Cells (UC-MSCs) for Treatment of Liver Failure
Brief Title: Safety and Efficacy of Human Mesenchymal Stem Cells for Treatment of Liver Failure
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Fu-Sheng Wang, Director, Beijing 302 Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Beijing302-003
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Liver Failure; Mesenchymal Stem Cells
Keywords: Liver Failure; Mesenchymal Stem Cells; Model for End-Stage Liver Disease; Ascite; Serum Albumin
MeSH Terms: conditions — Liver Failure | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional plus MSC treatment (Experimental): Participants will receive conventional treatment plus a dose of MSC from day 0 through the week 12 study visit. Participants will then be followed until 2 years study visit
  Interventions: Drug: Conventional plus MSC treatment
- Conventional plus pacebo treatment (Experimental): Participants will receive conventional plus placebo treatment from day 0 through the week 12 study visit. Participants will then be followed until 2 years study visit
  Interventions: Drug: Conventional plus pacebo treatment

INTERVENTIONS:
Drug: Conventional plus MSC treatment — Participants received conventional treatment and taken i.v., once per 4 week, at a dose of 0.5*10E6 MSC/kg body for 12 weeks.
  Arms: Conventional plus MSC treatment
Drug: Conventional plus pacebo treatment — Participants received conventional treatment and taken i.v., once per 4 week, at 50 ml saline for 12 weeks.
  Arms: Conventional plus pacebo treatment

SUMMARY:
Liver failure (LF) is a dramatic clinical syndrome with massive necrosis of liver cells. and liver transplantation is the only available therapeutic option for patients suffering with this condition. However, lack of donors, surgical complications, rejection, and high cost are serious problems. Previous study showed that bone marrow derived mesenchymal stem cells (BM-MSCs) replace hepatocytes in injured liver, and effectively rescue experimental liver failure and contribute to liver regeneration. In this study, the patients with LF will undergo administration of human umbilical cord mesenchymal stem cells (UC-MSCs) via peripheral vein transfusion to evaluate the safty and efficacy of UC-MSCs treatment for these patients.

DETAILED DESCRIPTION:
Liver failure (LF) is a severe life-threatening condition, and is a dramatic clinical syndrome with massive necrosis of liver cells, and liver transplantation is the only available therapeutic option for patients suffering with this condition. However, lack of donors, surgical complications, rejection, and high cost are serious problems. Since current therapeutic options for LF that is usually with extremely poor prognosis are still limited, recent studies indicate that mesenchymal stem cells (MSCs), due to their function in immune modulation and liver-damage repair, are of great therapeutic potential for this disease. Previous study showed that bone marrow derived mesenchymal stem cells (BM-MSCs) replace hepatocytes in injured liver, and effectively rescue experimental liver failure and contribute to liver regeneration.The purpose of this study is to investigate the safety and initial efficacy of human umbilical cord MSC (UC-MSCs) treatment for patients with LF. In this study, MSCs were isolated from umbilical cord and generated in appropriate growth medium. 50 LF patients with LF received i.v. transfusion of 0.5-1.0×106 cells/kg of MSCs as the treated group and other 20 LF patients with LF were transfused with placebo without MSCs as control group. All 70 of them received the routine management for liver failure. During the 2-year follow up, the evaluation of safty and efficacy will be undergone to help to establish innovative cell-based therapies for the treatment of diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years
2. Liver failure
3. Negative pregnancy test (female patients in fertile age)
4. Written consent

Exclusion Criteria:

1. Hepatocellular carcinoma or other malignancies
2. Severe problems in other vital organs(e.g.the heart,renal or lungs)
3. Pregnant or lactating women
4. Severe bacteria infection
5. Anticipated with difficulty of follow-up observation
6. Other candidates who are judged to be not applicable to this study by doctors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
The levels of serum Total Protein and Albumin | 2 years after treatment

SECONDARY OUTCOMES:
The levels of serum Total Bilirubin and Direct Bilirubin | 2 years after treatment
The levels of serum Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) and Cholinesterase (CHE) | 2 years after treatment
The level of alpha-fetoprotein (AFP) | 2 years after treatment
The content of ascites | 2 years after treatment
Survival rate and time | 2 years after treatment
Body temperature, tetter and allergy | Between 0 to 24 hours after UC-MSCs transfusion
The levels of Prothrombin Activity (PA) and Prothrombin Time (PT) | 2 years after treatment
The score for Model for End-Stage Liver Disease | 2 years after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, Professor, Principal Investigator — Beijing 302 Hospital
Locations (1):
- Beijing 302 Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Kuo TK, Hung SP, Chuang CH, Chen CT, Shih YR, Fang SC, Yang VW, Lee OK. Stem cell therapy for liver disease: parameters governing the success of using bone marrow mesenchymal stem cells. Gastroenterology. 2008 Jun;134(7):2111-21, 2121.e1-3. doi: 10.1053/j.gastro.2008.03.015. Epub 2008 Mar 12. PMID 18455168
- [Background] Campard D, Lysy PA, Najimi M, Sokal EM. Native umbilical cord matrix stem cells express hepatic markers and differentiate into hepatocyte-like cells. Gastroenterology. 2008 Mar;134(3):833-48. doi: 10.1053/j.gastro.2007.12.024. Epub 2007 Dec 23. PMID 18243183
- [Background] Terai S, Ishikawa T, Omori K, Aoyama K, Marumoto Y, Urata Y, Yokoyama Y, Uchida K, Yamasaki T, Fujii Y, Okita K, Sakaida I. Improved liver function in patients with liver cirrhosis after autologous bone marrow cell infusion therapy. Stem Cells. 2006 Oct;24(10):2292-8. doi: 10.1634/stemcells.2005-0542. Epub 2006 Jun 15. PMID 16778155
- [Result] Mohamadnejad M, Alimoghaddam K, Mohyeddin-Bonab M, Bagheri M, Bashtar M, Ghanaati H, Baharvand H, Ghavamzadeh A, Malekzadeh R. Phase 1 trial of autologous bone marrow mesenchymal stem cell transplantation in patients with decompensated liver cirrhosis. Arch Iran Med. 2007 Oct;10(4):459-66. PMID 17903050
- [Result] Kharaziha P, Hellstrom PM, Noorinayer B, Farzaneh F, Aghajani K, Jafari F, Telkabadi M, Atashi A, Honardoost M, Zali MR, Soleimani M. Improvement of liver function in liver cirrhosis patients after autologous mesenchymal stem cell injection: a phase I-II clinical trial. Eur J Gastroenterol Hepatol. 2009 Oct;21(10):1199-205. doi: 10.1097/MEG.0b013e32832a1f6c. PMID 19455046